CLINICAL TRIAL: NCT04189614
Title: A Phase 1b Efficacy and Safety Study of Cofetuzumab Pelidotin (ABBV-647, a PTK7-Targeting Antibody Drug Conjugate) in Subjects With PTK7-Expressing, Recurrent Non-Small Cell Lung Cancer
Brief Title: An Efficacy and Safety Study of Cofetuzumab Pelidotin in Participants With PTK7-Expressing, Recurrent Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-611; 2019-003472-39 (EudraCT Number)
Record Dates: First submitted 2019-12-05; First posted 2019-12-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small Cell Lung Cancer (NCSLC); PTK7-Expressing Tumor; Antibody Drug Conjugate; cofetuzumab pelidotin; ABBV-647; Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — cofetuzumab pelidotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cofetuzumab Pelidotin (Experimental): Participants will receive 2.8mg/kg of cofetuzumab pelidotin by IV every 3 weeks
  Interventions: Drug: Cofetuzumab Pelidotin

INTERVENTIONS:
Drug: Cofetuzumab Pelidotin — Intravenous (IV) infusion
  Other Names: ABBV-647

SUMMARY:
This study is being done to determine the efficacy and safety of cofetuzumab pelidotin in the PTK7-expressing, recurrent non-small cell lung cancer (NSCLC) population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC) with PTK7-expressing tumor using an immunohistochemistry (IHC) assay previously validated at a designated laboratory
* Recurrent NSCLC that has progressed after treatment with at least the following approved therapies with demonstrated clinical benefit: a platinum-based chemotherapy doublet and an immune checkpoint inhibitor for tumors without targetable genetic alterations; a platinum-based chemotherapy doublet and targeted agent(s) for tumors with targeted genetic alterations
* Received ≤ 2 prior lines of systemic therapy, including no more than 1 line of systemic cytotoxic chemotherapy (≤ 3 prior lines for tumors treated with targeted agent(s) for genetic alterations, including no more than 1 line of systemic chemotherapy)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Adequate bone marrow, renal, and hepatic function per the protocol

Exclusion Criteria:

* Known uncontrolled metastases to the central nervous system (CNS). Participants with CNS metastases may be eligible provided that definitive therapy has been given, and participants are asymptomatic and off systemic steroids and anticonvulsants used for management of brain metastases for at least 2 weeks prior to the first dose of study drug
* Unresolved clinically significant adverse events Grade ≥ 2 from prior anticancer therapy (with the exception of alopecia or anemia)
* Has clinically significant medical condition(s) as described in the protocol
* Received anticancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 28 days prior to the first dose of study drug (no washout period required for participants on EGFR tyrosine kinase inhibitors). Palliative radiation therapy for bone, skin or subcutaneous metastases with 10 fractions or less is not subject to a washout period
* Received anti-cancer herbal therapies within 7 days prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria and defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from the participant's initial response (CR or PR) to the first occurrence of radiographic progression or death from any cause.
Progression Free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from the participant's first dose of study drug until radiographic progression or death from any cause.
Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from the participant's first dose of study drug until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (12):
  - University of Alabama at Birmingham - Main /ID# 213605, Birmingham, Alabama
  - Highlands Oncology Group, PA /ID# 215383, Springdale, Arkansas
  - Duplicate_Stanford University School of Med /ID# 213450, Stanford, California
  - Univ of Colorado Cancer Center /ID# 215295, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center /ID# 216433, Miami, Florida
  - Moffitt Cancer Center /ID# 215101, Tampa, Florida
  - Washington University-School of Medicine /ID# 213453, St Louis, Missouri
  - The Ohio State University /ID# 211088, Columbus, Ohio
  - Tennessee Oncology, PLLC /ID# 215326, Nashville, Tennessee
  - Oncology Consultants /ID# 215932, Houston, Texas
  - University of Texas MD Anderson Cancer Center /ID# 215876, Houston, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 216427, Fairfax, Virginia
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 217538, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 217536, Haifa
  - Rabin Medical Center /ID# 217537, Petah Tikva
- Japan (2):
  - National Cancer Center Hospital East /ID# 218537, Kashiwa-shi, Chiba
  - National Cancer Center Hospital /ID# 218536, Chuo-ku, Tokyo
- South Korea (4):
  - CHA Bundang Medical Center /ID# 232514, Seongnam, Gyeonggido
  - Asan Medical Center /ID# 222280, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 222906, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 222281, Seoul
- Spain (3):
  - Hospital Universitario Vall d'Hebron /ID# 215729, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 215110, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 215102, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital /ID# 222602, Tainan
  - Linkou Chang Gung Memorial Hospital /ID# 222603, Taoyuan

IPD SHARING:
Plan to Share IPD: No